CLINICAL TRIAL: NCT04033523
Title: High-Intensity Interval Training Recuperates Capacity of Endogenous Thrombin Generation in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, PhD, Rehabilitation Science, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201301077A3
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; High-intensity Interval Training
Keywords: heart failure; exercise; microparticles; thrombin
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity-interval training (HIIT) (Experimental): The HF group performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 3 days/week for 12 weeks
  Interventions: Behavioral: HIIT
- normal counterparts (No Intervention): gender-matched normal counterparts (NC) did not receive any form of intervention

INTERVENTIONS:
Behavioral: HIIT — The HF group performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 3 days/week for 12 weeks
  Arms: High intensity-interval training (HIIT)

SUMMARY:
Consumptive coagulopathy is associated with increased mortality in patients with heart failure (HF). Physical activity influences the risk of major vascular thrombotic events. This study investigates how high-intensity interval training (HIIT) affects the capacity of endogenous thrombin generation (TG) by modulating circulatory procoagulant microparticles (MPs) in HF patients. Thirty-eight HF patients and 38 age- and gender-matched normal counterparts (NC) were recruited into this study. The HF group performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 3 days/week for 12 weeks, whereas the NC group did not receive any form of intervention. Plasma TG kinetics, procoagulant MPs, coagulation-related factors, and oxidative stress/proinflammatory status were analyzed. The results demonstrated that the HF group exhibited (i) less endogenous thrombin potential (ETP) and TG rate, (ii) lower concentration/activity of tissue factor (TF) and counts of TF-rich MPs derived from blood cells, and (iiii) higher vascular endothelial shedding and plasma myeloperoxidase and interleukin-6 concentrations, compared to the NC group did. However, HIIT elevated plasma ETP and TG rate, as well as, TF concentration/activity and blood cell-derived procoagulant MP levels in the HF patients. Moreover, the exercise regimen also decreased vascular endothelial shedding and plasma myeloperoxidase and interleukin-6 concentrations in patients with HF. Hence, we conclude that HF reduces the capacity of endogenous TG in plasma, which is associated with decreased (or consumed) circulatory procoagulant MP levels. However, HIIT alleviates HF-declined endogenous TG capacity and vascular endothelial damage through recuperating TF-related coagulation activity and suppressing oxidative stress/proinflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* The HF was diagnosed if the patients had a left ventricular ejection fraction (LVEF) <40%.
* All HF patients were New York Heart Association (NYHA) functional class II or III and had received optimal treatment for at least 12 months according to American Heart Association/American College of Cardiology guidelines.

Exclusion Criteria:

* Patients with the presence of atrial fibrillation/flutter, second/third degree heart block, history of life-threatening ventricular arrhythmias, recent unstable angina, myocardial infarction or coronary revascularization (<4 weeks), uncontrolled diabetes mellitus, severe chronic obstructive pulmonary disease, or symptomatic cerebral vascular disease within 12 months, collagen vascular disease, alcohol or drug abuse during the previous 12 months or significant renal or hepatic disease were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Microparticles derived from blood cells and shedding endothelial cells | 12 weeks
  Platelet-poor plasma (PPP) was separated from whole blood by centrifugation at 1,600g for 10 min at room temperature.
  The quantification of microparticles in PPP was determined by a three-color FACScan flow cytometer.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 12 weeks
  evaluate cardiac hemodynamic response to exercise by noninvasive continuous cardiac output monitoring system

OTHER OUTCOMES:
Thrombin generation assay | 12 weeks
  PPP was measure the rate of thrombin generation using the calibrated automated thrombogram (CAT) assay (Synapse/Thrombinoscope BV).